CLINICAL TRIAL: NCT02485249
Title: Open-label, Multli-center, Phase 1b/2a Clinical Trial Designed to Evaluate the Safety and Efficacy of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution in Patients With Macular Edema
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGP-437-007
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Macular Edema
Keywords: Iontophoresis; Macular Edema; Ophthalmology
MeSH Terms: conditions — Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexamethasone Phosphate (Experimental): Dexamethasone Phosphate Ophthalmic solution (40 mg/mL) delivered by ocular iontophoresis consisting of 14.0 mA-min at 3.5 mA on Day 0, Day 4, and Day 14
  Interventions: Drug: Dexamethasone Phosphate Ophthalmic

INTERVENTIONS:
Drug: Dexamethasone Phosphate Ophthalmic — Transscleral iontophoresis delivery of EGP-437 (dexamethasone phosphate formulated for ocular iontophoresis)
  Other Names: 40 mg/mL Dexamethasone Phosphate Ophthalmic

SUMMARY:
To evaluate the safety and efficacy of ocular iontophoresis with dexamethasone phosphate ophthalmic solution, EGP-437, using the EyeGate® II Drug Delivery System (EGDS) in patients with macular edema (ME)

DETAILED DESCRIPTION:
This will be a Phase 1b/2a, exploratory, open-label study, in which up to 20 eligible ME patients will be enrolled at up to 5 clinical sites in the U.S. Twenty eyes of 20 patients will be enrolled which means that only one eye will be treated with study treatment in patients who present at Visit 1 with bilateral ME. In situations where both eyes of a patient are eligible for the study, the eye with the shorter duration of ME will be the study eye.9 The investigator will designate the study eye when both eligible eyes have been diagnosed with ME at the same time. Potential patients who are interested in participating in the study will be provided an informed consent form (ICF) prior to screening. Patient eligibility will be assessed at Visit 1 (Day 0), the baseline visit, by spectral SD-OCT and measurement of IOP, in addition to review of the patient's medical and ophthalmic history and recent concomitant medications history. Study Treatment will be administered on Day 0, Day 4, and Day 9 (Visits 1, 2, and 3). Subjects will be scheduled to return to the clinic for post-treatment assessments during Visits 4 and 5 (Day 14 and Day 21 or Day 28).

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 to 90 years 2. Have diagnosis of ME secondary to one of the following diagnosed conditions:

  1. Central or branch retinal vein occlusion (CRVO or BRVO) with a mean CST ≥ 300µm on SD-OCT images taken at the baseline visit (Day 0)
  2. Diabetic macular edema (DME) with a mean CST ≥ 300µm on SD-OCT images taken at the baseline visit (Day 0)
  3. Cystoid macular edema (CME) secondary to having undergone a previous PPV and having a mean CST ≥ 300µm on SD-OCT images taken at the baseline visit (Day 0) having a history of previous positive response to steroid treatment 3. Receive, understand, and sign a copy of the ICF 4. Be able to return for all study visits and willing to comply with all study related instructions

     Exclusion Criteria:

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Anatomic improvement measured as reduction in mean central subfield thickness as evaluated by spectral-domain-optical coherence tomography | Day 4, Day 9, Day 14, and Day 21

SECONDARY OUTCOMES:
Changes in macular volume as evaluated by spectral-domain-optical coherence tomography | Day 4, Day 9, Day 14, and Day 21
Qualitative review of spectral-domain-optical coherence tomography scans | Day 4, Day 9, Day 14, and Day 21
Dilated fundus exam | Day 4, Day 9, Day 14, and Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Brandano, Study Director — EyeGate
Locations (1):
- Ophthalmic Consultants of Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided